CLINICAL TRIAL: NCT02842320
Title: Targeting Leukemic Stem Cell Expressing the IL-1RAP Protein in Chronic Myelogenous Leukemia (CML)
Acronym: CAR-LMC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P/2015/244
Record Dates: First submitted 2016-07-20; First posted 2016-07-22 (Estimated); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Additional biological samples (Experimental): Bone marrow sample and blood collected at J0 (screening visit), and at 3, 6, 12, 18 and 24 months and at each additional consultations (relapse ...)
  Interventions: Other: biological samples

INTERVENTIONS:
Other: biological samples — bone marrow and blood

SUMMARY:
The tyrosine kinase inhibitor therapy (iTKs) is the first-line treatment of chronic myelogenous leukemia (CML).

Its effectiveness in controlling the progression of the disease is such that it is possible today to consider stopping treatment in patients with deep molecular response (> RM4.0).

Only in about 50% of cases, patients relapse. It has been shown in these patients that hematopoietic stem cells (HSCs) are persistant, quiescent and insensitive to iTKs. These cells are probably at the origin of relapse. It is therefore necessary to develop complementary therapies to cure the disease and consider discontinuation iTKs The development of anti-tumor immunotherapy approach using genetically modified T cells to express a chimeric antigen receptor (CAR) and specifically targeting CML CSH + could address this issue. The membrane expression of the IL-1-RAP protein could be an interesting target.

ELIGIBILITY:
Inclusion Criteria:

* patients for whom there is a strong suspicion of CML diagnosed as part of routine activity.
* written informed consent

Exclusion Criteria:

* patient with atypical CML
* patient with a non SMP CML
* patients previously treated with interferon
* patient enrolled in another study therapy or within the exclusion period thereof
* pregnant or breast-feeding women
* patient under guardianship, curator or under the protection of justice.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2015-10-14 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
IL1RAP protein expression on the surface of cells detected by flow cytometry | up to 2 years after inclusion

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Hôpital Nord Franche-Comté, Belfort
  - Centre Hospitalier Régional Universitaire de Besançon, Besançon
  - CHU de Dijon, Dijon
  - CHI de Haute-Saône, Vesoul

IPD SHARING:
Plan to Share IPD: No